CLINICAL TRIAL: NCT03488160
Title: CAR-T Cell Therapy for Relapsed / Refractory CD19 Positive Clinical Study on the Safety and Effectiveness of Lymphoma
Brief Title: CAR-T Treatment for Relapse / Refractory Type Safety and Effectiveness of Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinobioway Cell Therapy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sinobiowayCT
Record Dates: First submitted 2018-03-26; First posted 2018-04-04 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Lymphoma
Keywords: lymphoma CAR-T
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) Dosage form：injection Dosage:100ml/time Frequency:the first day,the second day Duration:total two times
  Interventions: Biological: CD19-targeted CAR-T cells

INTERVENTIONS:
Biological: CD19-targeted CAR-T cells — This study have only one arm that is CAR-T experimental arm. Firstly all participators will be attended the screening, who passed the screening for the treatment of CAR-T cells, the CAR-CD19-modified T cells can recognize and kill tumor cells in the body，follow-up 35 months..

SUMMARY:
The safety and feasibility of CAR-T cells (CD19.CAR-T) targeted at CD19 in the treatment of relapsed / refractory CD19 positive lymphoma were determined, and the proliferation and survival time of CD19.CAR-T cells in patients were determined.

DETAILED DESCRIPTION:
The sponsors of this research also studied CD19.CAR-T cells for the treatment of leukemia and lymphoma, two courses of three transfusion 14 days after infection process standard training program , the safety and effectiveness have accumulated some of the data. In this study, the investigators will regenerate the cultured cells for 2 times in a course of treatment, and enter the patient's body . The investigators observed the safety and efficacy of CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 16 years old, less than 70 years old, sex is not limited, race is not limited;
2. The pathological diagnosis was CD19 positive expression of B type lymphoma relapsed / refractory, meet any one of the following can be diagnosed with relapsed / refractory lymphoma: 1）the standard scheme of standardized treatment of more than 4 courses in 50%, or the condition of tumor size;2） standard treatment of CR, but the recurrence of use the original scheme or the current national consensus recommended second-line treatment can not get CR again;3） the relapse after haematopoietic stem cell transplantation;
3. The patient needs to have a lesion that can be used to detect or evaluate the disease.
4. 0~1 score of physical status score of the eastern cancer cooperation group (ECOG).
5. At the time of collection of peripheral white blood cell counts over 1 * 10^9/L;
6. Expected survival time > 90 days;
7. Patients have the ability to know and sign informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Uncontrolled infection;
3. HIV infected people, hepatitis B or HCV active stage;
4. Needs patients with long-term immunosuppressive therapy (such as allergies, autoimmune diseases, GVHD, etc.).
5. Combined with active central nervous system malignant tumor invading;
6. Has abnormal coagulation function, and there are patients with serious thrombus.
7. Organ failure (Appendix); A. heart: Grade II and above; B. liver: higher than grade II; C. kidney: second stages of renal insufficiency and above; D. lung: the second grade was slightly hypofunction and above. E. brain: metastatic or active lesion of the central nervous system.
8. Patients who participated in other clinical trials in the past 30 days or in other clinical trials;
9. Researchers believe that patients are not suitable for the study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-04-10 (Estimated); Primary Completion 2019-04-10 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: The overall efficiency | [Time Frame: 3 years]
  Complete remission (CR) number+The number of partial response (PR)/Total number of cases being treated

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wu, Principal Investigator — Investigator associate chief physician; Kaiyang Ding, Principal Investigator — Chief physician
Locations (1):
- The west area of the First Affiliated Hospital of University of Science & Technology China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No